CLINICAL TRIAL: NCT01782014
Title: Water Infusion and Carbon Dioxide Insufflation Versus Air Insufflation Versus Air Insufflation Techniques in Screening Colonoscopies in the United States: A Comparative Study Evaluating Safety, Efficacy and Adenoma Detection Rate (ADR)
Brief Title: Comparison of Adenoma Detection Rate Among Water, Carbon Dioxide and Air Methods of Minimal Sedation Colonoscopy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 5130003; LLUMCGI2013 (Other: Loma Linda University)
Record Dates: First submitted 2013-01-27; First posted 2013-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2014-09

CONDITIONS: Screening Colonoscopy
Keywords: Screening colonoscopy; Water method; Carbon dioxide method; Air method; Water versus carbon dioxide versus air insufflation colonoscopy; Adenoma Detection Rate; Pain Scores in colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Water Insufflation (Experimental): Colonoscopy using water insufflation
  Interventions: Procedure: colonoscopy
- Carbon dioxide insufflation (Active Comparator): Colonoscopy using carbon dioxide insufflation
  Interventions: Procedure: colonoscopy
- Air insufflation (Active Comparator): Colonoscopy using air insufflation
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — colonoscopy using different methods of insufflation

SUMMARY:
The purpose of this study is to determine which of the methods of colonoscopy viz. water insufflation or air insufflation or carbon dioxide insufflation is better in detecting the adenomas in colon and also which of these methods is best tolerated by patients.

Hypothesis: the investigators hypothesize that in patients undergoing first time screening colonoscopy a higher Adenoma Detection Rate will be found in the proximal colon in the group randomized to the water method compared to those randomized to the air or CO2 insufflation methods

DETAILED DESCRIPTION:
Significance:

ADR is an independent predictor of risk of post screening colonoscopy colon cancer. A simple method solely controlled by the colonoscopist that enhances proximal ADR holds the promise of rectifying some of the unresolved shortcomings of screening colonoscopy in failing to reduce the occurrence of post screening incident cancers in the proximal colon and the associated cancer mortality.

Hypotheses & Specific Aims:

Primary Hypothesis:

In patients undergoing first time screening a higher ADR will be found in the proximal colon in those randomized to the water method compared to those randomized to the air method or CO2 method.

Secondary Hypotheses:

The examination method but not co-variables, procedure-related or patient-centered outcomes, is an independent predictor of proximal colon ADR.

Specific Aims:

This is a prospective, randomized, single-blinded controlled study to compare the study (water) and control 1 (air) method and control 2 (CO2 method) to aid insertion of the colonoscope. The proximal colon ADR, total ADR, co-variables, procedure-related and patient-centered outcomes and adverse event during and within 30 days of colonoscopy will be recorded and compared between the study and control methods.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients with average risk for colorectal cancer, who are scheduled for first-time screening colonoscopy, will be enrolled.

Exclusion Criteria:

* decline to be randomized
* unable to give consent
* non-screening (surveillance or diagnostic) colonoscopy
* current participation in other colonoscopy studies
* a medical condition that could increase the risk associated with colonoscopy
* pregnancy
* those with a known family history of polyposis syndromes or a family history of colon cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate, proximal colon and total | Day 1, At time of colonoscopy
  The number of adenomas detected in proximal colon and total number of adenomas detected during the procedure will be compared between the three methods

SECONDARY OUTCOMES:
Pain scores | during and immediately after colonoscopy on day 1
  Visual Analog Scales will be used to calculate the pain scores based on the discomfort/pain experienced by the patient
Sedation requirements | Collected at Day 1, during the procedure
  The amount of sedation required to complete the patient's colonoscopy.

OTHER OUTCOMES:
Patient overall satisfaction score | immediately after colonoscopy on day 1
  patient satisfaction will be scored on a Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kendrick Che, DO, Principal Investigator — Loma Linda University Medical Center; Terrence Lewis, MD, Study Chair — Loma Linda University Medical Center; Michael Walter, MD, Study Chair — Loma Linda University Medical Center
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

REFERENCES:
- [Result] Leung FW, Aharonian HS, Leung JW, Guth PH, Jackson G. Impact of a novel water method on scheduled unsedated colonoscopy in U.S. veterans. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):546-50. doi: 10.1016/j.gie.2008.08.014. PMID 19231497
- [Result] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Result] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Result] Leung JW, Do LD, Siao-Salera RM, Ngo C, Parikh DA, Mann SK, Leung FW. Retrospective analysis showing the water method increased adenoma detection rate - a hypothesis generating observation. J Interv Gastroenterol. 2011 Jan;1(1):3-7. doi: 10.4161/jig.1.1.14585. PMID 21686105
- [Result] Leung FW, Leung JW, Siao-Salera RM, Mann SK. The water method significantly enhances proximal diminutive adenoma detection rate in unsedated patients. J Interv Gastroenterol. 2011 Jan;1(1):8-13. doi: 10.4161/jig.1.1.14587. PMID 21686106
- [Result] Leung FW, Leung JW, Siao-Salera RM, Mann SK, Jackson G. The water method significantly enhances detection of diminutive lesions (adenoma and hyperplastic polyp combined) in the proximal colon in screening colonoscopy - data derived from two RCT in US veterans. J Interv Gastroenterol. 2011 Apr;1(2):48-52. doi: 10.4161/jig.1.2.16826. PMID 21776425
- [Result] Stevenson GW, Wilson JA, Wilkinson J, Norman G, Goodacre RL. Pain following colonoscopy: elimination with carbon dioxide. Gastrointest Endosc. 1992 Sep-Oct;38(5):564-7. doi: 10.1016/s0016-5107(92)70517-3. PMID 1397911
- [Result] Wong JC, Yau KK, Cheung HY, Wong DC, Chung CC, Li MK. Towards painless colonoscopy: a randomized controlled trial on carbon dioxide-insufflating colonoscopy. ANZ J Surg. 2008 Oct;78(10):871-4. doi: 10.1111/j.1445-2197.2008.04683.x. PMID 18959640
- [Result] Leung FW, Leung JW, Mann SK, Friedland S, Ramirez FC. The water method significantly enhances patient-centered outcomes in sedated and unsedated colonoscopy. Endoscopy. 2011 Sep;43(9):816-21. doi: 10.1055/s-0030-1256407. Epub 2011 May 24. PMID 21611947